CLINICAL TRIAL: NCT05892523
Title: Influence of Spinal Deformity on Acetabular Cup Position in THA.
Brief Title: Influence of Spinal Deformity on THA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Rahman Mazhar, Assistant lecturer, Assiut University
Other Study IDs: spinal deformity in THA
Record Dates: First submitted 2023-05-25; First posted 2023-06-07 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: THA
MeSH Terms: interventions — Tacrine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: THA — positioning the acetabular cup regarding abduction and anteversion angles with or without concern to spinal deformity

SUMMARY:
The aim of the study is to understand the effect of spinal deformity and altered sagittal plane parameters of lumbosacral complex on acetabular cup position in THA.

DETAILED DESCRIPTION:
Investigators will Find out if there is change in the acetabular cup including the abduction and anteversion angles in patients who had THA and has spinal deformity

ELIGIBILITY:
Inclusion Criteria:

* all patients who had primary THA in 6 month duration
* patients from 30 to 70 years old with primary THA

Exclusion Criteria:

* patients who have ankylosing spondylitis
* patients with revised THA
* patients with associated injuries in lower limb

Ages: 30 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients from 30 to 70 years old with primary THA and spinal deformity
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-11-08 (Estimated); Primary Completion 2024-11-08 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
change of acetabular cup position in spinal deformity | immediate post operative X-ray hip anteroposterior and cross table lateral views in supine position measuring cup abduction and anteversion angles and 3 month post operative X-ray hip and lumbosacral anteroposterior and lateral views in standing position
  change of acetabular cup abduction and anteversion angles in patients who has THA and spinal deformity

SECONDARY OUTCOMES:
complications of THA mainly hip dislocation and HOOS hip survey | 3 month duration post operatively
  post-operative hip dislocation

CONTACTS AND LOCATIONS:
Overall Officials: Hatem M Abdel-Moneim Bakr, professor, Study Chair — Assiut University

REFERENCES:
- [Background] Phan D, Bederman SS, Schwarzkopf R. The influence of sagittal spinal deformity on anteversion of the acetabular component in total hip arthroplasty. Bone Joint J. 2015 Aug;97-B(8):1017-23. doi: 10.1302/0301-620X.97B8.35700. PMID 26224815
- [Background] Blizzard DJ, Nickel BT, Seyler TM, Bolognesi MP. The Impact of Lumbar Spine Disease and Deformity on Total Hip Arthroplasty Outcomes. Orthop Clin North Am. 2016 Jan;47(1):19-28. doi: 10.1016/j.ocl.2015.08.005. PMID 26614917